CLINICAL TRIAL: NCT04665115
Title: A Prospective Study of Patients With B-Cell Hematologic Malignancies on Ibrutinib Therapy Who Are Infected With Coronavirus Disease 2019 (COVID-19)
Brief Title: Ibrutinib for the Treatment of Patients With B-Cell Malignancies Who Are Infected With Coronavirus Disease 2019 (COVID-19)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanently closed 11/19/201. The widespread availability of COVID vaccination, the projected decline in infection rates, and the increasing use of non-ibrutinib containing BTKi therapy, we have not been able to get support for this study
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-LY-2001; NCI-2020-11785 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-LY-2001 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Asymptomatic COVID-19 Infection Laboratory-Confirmed; B-Cell Neoplasm; Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma; Symptomatic COVID-19 Infection Laboratory-Confirmed; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort I (ibrutinib) (Experimental): Patients may continue to receive ibrutinib PO daily or stop ibrutinib per provider's discretion.
  Interventions: Drug: Ibrutinib; Other: Quality-of-Life Assessment
- Cohort II Arm 2A (ibrutinib) (Experimental): Patients continue to receive ibrutinib PO daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Quality-of-Life Assessment
- Cohort II Arm 2B (temporary interruption) (Experimental): Patients undergo temporary interruption of ibrutinib for up to 28 days unless they are discharged home and are thought to be medically fit by the primary caregiver to resume therapy according to their primary treating oncologist.
  Interventions: Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
  Arms: Cohort I (ibrutinib); Cohort II Arm 2A (ibrutinib)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the effects of ibrutinib in treating patients with B-cell malignancies who are infected with COVID-19. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Ibrutinib is a first in class Bruton tyrosine kinase inhibitor (BTKi), for the treatment of B-cell malignancies. This study is being done to determine if taking ibrutinib after contracting COVID-19 will make symptoms better or worse.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize and describe the patterns of temporary interruption vs. continuation of ibrutinib after their coronavirus disease 2019 (COVID-19) diagnosis and their corresponding rates of hospitalization and/or death by day 28 in an observational cohort of COVID-19 infected patients treated with ibrutinib therapy as their standard of care. (Cohort 1) II. To determine if continuation of ibrutinib during COVID-19 infection among patients who are hospitalized can result in decreased need for mechanical ventilation and decreased mortality by day 28 compared to patients who suspend temporarily ibrutinib treatment after their COVID-19 diagnosis. (Cohort 2)

SECONDARY OBJECTIVES I. To determine the average length of time from diagnosis of COVID-19 infection to need for hospitalization due to worsening disease. (Cohort 1) II. To determine the rate of viral clearance on days 15, 28, 42, and 56 after registration. (Cohort 1) III. To evaluate coagulation parameters at baseline, and on days 15 and 28 after registration. (Cohort 1) IV. To determine the incidence of arterial and venous thrombosis as well as bleeding complications. (Cohort 1) V. To evaluate patient-reported health status and quality of life using the patient reported outcome (PRO)-Common Terminology Criteria for Adverse Events (CTCAE). (Cohort 1) VI. To determine if patients develop a "flare phenomenon" if ibrutinib is stopped. (Cohort 1) VII. To evaluate the patterns and timing of restarting ibrutinib in those patients who suspended their ibrutinib treatment after their COVID-19 diagnosis. (Cohort 1) VIII. To evaluate the association of patient outcomes stratified by the Charlson Co-morbidity index (CCI). (Cohort 1) IX. To evaluate the safety and tolerability of continuation of ibrutinib. (Cohort 1) X. To evaluate if continued treatment with ibrutinib can reduce the proportion of patients who die due to any cause in the 28 days after randomization compared to patients who stop ibrutinib in COVID-19 positive patients who are hospitalized at the time of study enrollment. (Cohort 2) XI. To evaluate the incidence of mechanical ventilation in hospitalized patients, and whether continued ibrutinib therapy reduces this incidence compared to stopping ibrutinib. (Cohort 2) XII. To determine whether continued ibrutinib can significantly improve the viral clearance rate at baseline, and on days 8, 15, 28, 42 and 56 days after randomization compared to those who temporarily interrupt ibrutinib. (Cohort 2) XIII. To evaluate coagulation parameters at baseline, and on days 8, 15, and 28 after randomization among patients who continue ibrutinib compared to those who discontinue ibrutinib. (Cohort 2) XIV. To determine the incidence of arterial and venous thrombosis as well as bleeding complications in patients who continue ibrutinib compared to those who stop it. (Cohort 2) XV. To determine if patients who are randomized to stopping ibrutinib develop "flare phenomenon". (Cohort 2) XVI. To evaluate the association of patient outcomes stratified by the Charlson Co-morbidity index (CCI). (Cohort 2)

CORRELATIVE RESEARCH OBJECTIVES:

I. To evaluate the association of inflammatory status with COVID severity. II. To determine the proportion of patients who develop antibodies to SARS-CoV2, especially given that patients with B cell malignancies tend to have inadequate responses to vaccines and often suffer from hypogammaglobulinemia.

III. To determine changes in the immune profile by advanced flow cytometry given that the status of the immune system , both innate and adaptive , may dictate ultimate host management and clearance of COVID infections.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients may continue to receive ibrutinib orally (PO) daily or stop ibrutinib per provider's discretion.

COHORT II: Patients are randomized to 1 of 2 arms.

ARM 2A: Patients continue to receive ibrutinib PO daily in the absence of disease progression or unacceptable toxicity.

ARM 2B: Patients undergo temporary interruption of ibrutinib for up to 28 days unless they are discharged home and are thought to be medically fit by the primary caregiver to resume therapy according to their primary treating oncologist.

After completion of study treatment, patients are followed up at 42, 56, and 84 days.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION INCLUSION
* (COHORT 1): Age >= 18 years
* COHORT 1: Laboratory confirmed diagnosis of COVID-19 through confirmation of SARS-Co-V2 via reverse transcriptase polymerase chain reaction (RT-PCR) or any Food and Drug Administration (FDA) approved method. The date of test result is required to be =< 7 days prior to registration (NOTE: please use the date the test was resulted and NOT the date when the test was collected)
* COHORT 1: Patient is on ibrutinib for the following approved FDA indications, including:

  * Chronic lymphocytic leukemia/Small lymphocytic lymphoma
  * Mantle cell lymphoma
  * Waldenstrom macroglobulinemia
  * Marginal zone lymphoma
* COHORT 1: Patients have been on standard dose ibrutinib therapy (420 mg daily for chronic lymphocytic leukemia [CLL]/small lymphocytic lymphoma [SLL] and Waldenstrom/Waldenstrom macroglobulinemia, and 560 mg daily for mantle cell lymphoma and marginal zone lymphoma) for at least 6 months prior to diagnosis of COVID-19 infection; and there is no evidence of disease progression of the primary malignancy for which ibrutinib is being used

  * NOTE: Patients are allowed to receive standard treatment as per local institutional guidelines for the treatment of COVID-19 at the same time the patient is enrolled on this trial
* COHORT 1: Provide informed written consent =< 7 days prior to registration
* COHORT 1: Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: During the active monitoring phase of a study (i.e., active treatment and clinical follow-up), participants must be willing to return to the consenting institution for follow-up. All of these visits will be virtual (phone or video) ONLY
* COHORT 1: Willing to provide blood specimens for correlative research purposes
* RANDOMIZATION INCLUSION
* COHORT 2: Age >= 18 years
* COHORT 2: Laboratory confirmed diagnosis of COVID-19 through confirmation of SARS-Co-V2 via RT-PCR or any FDA approved method. The date of test result is required to be =< 7 days prior to registration (NOTE: please use the date the test was resulted and NOT the date when the test was collected)
* COHORT 2: Patient is on ibrutinib for the following approved FDA indications, including:

  * Chronic lymphocytic leukemia/Small lymphocytic lymphoma
  * Mantle cell lymphoma
  * Waldenstrom macroglobulinemia
  * Marginal zone lymphoma
* COHORT 2: Patients have been on standard dose ibrutinib therapy (420 mg daily for CLL/SLL and Waldenstrom macroglobulinemia, and 560 mg daily for mantle cell lymphoma and marginal zone lymphoma) for at least 6 months prior to diagnosis of COVID-19 infection; and there is no evidence of disease progression of the primary malignancy for which ibrutinib is being used

  * NOTE: Patients are allowed to receive standard treatment as per local institutional guidelines for the treatment of COVID-19 at the same time the patient is enrolled on this trial
* COHORT 2: Provide informed written consent =< 7 days prior to registration
* COHORT 2: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

  * Note: During the Active Monitoring Phase of a study (i.e., active treatment and clinical follow-up), participants must be willing to return to the consenting institution for follow-up. All of these visits will be virtual (phone or video) ONLY
* COHORT 2: Willing to provide blood specimens for correlative research purposes
* COHORT 2: Absolute neutrophil count (ANC) > 750 cells/mm^3 (0.75 x 10^9/L)
* COHORT 2: Platelet count > 50,000 cells/mm^3 (50 x 10^9/L)
* COHORT 2: Estimated creatinine clearance (CrCl) >= 30 mL/min (Cockcroft-Gault)
* COHORT 2: Bilirubin =< 2.0 x upper limit of normal (ULN) (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* COHORT 2: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 5 x ULN
* COHORT 2: Prothrombin time (PT)/International normal ratio (INR) < 1.5 x (upper limit of normal) ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder)

Exclusion Criteria:

* REGISTRATION EXCLUSION
* COHORT 1: Patient is receiving ibrutinib therapy for chronic graft-versus-host disease (cGVHD)
* COHORT 1: Patient is currently receiving (or has in the past 6 months) another treatment in combination with ibrutinib, such as anti-CD20 monoclonal antibody, BCL-2 antagonists such as venetoclax, or other novel treatments or chemotherapeutic agents. For clarification regarding specific medications not listed here, please discuss with the principal investigator
* COHORT 1: Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon) within 7 days of first dose of study drug and while on study
* COHORT 1: Concomitant use of a strong CYP3A inhibitor
* COHORT 1: Vaccinated with a live, attenuated vaccine within 4 weeks
* COHORT 1: Patients with chronic liver disease and hepatic impairment meeting Child Pugh class C
* COHORT 1: History of stroke or intracranial hemorrhage within 6 months before registration
* COHORT 1: History of bleeding diathesis (e.g. hemophilia, von Willebrand/Waldenstrom disease)
* COHORT 1: Clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to registration
* COHORT 1: Chemotherapy for other malignancies
* COHORT 1: Concurrent systemic immunosuppressant therapy within 21 days of the first dose of study drug with the exception of that which is part of the standard of care for COVID-19
* COHORT 1: Major surgery within 4 weeks of registration
* COHORT 1: Female subjects who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or within 1 month of last dose of study drug. Male subjects who plan to father a child while enrolled in this study or within 3 months after the last dose of study drug
* RANDOMIZATION EXCLUSION
* COHORT 2: Patient is receiving ibrutinib on a clinical trial for their underlying B-cell malignancy
* COHORT 2: Patient is receiving ibrutinib therapy for chronic graft-versus-host disease (cGVHD)
* COHORT 2: Patient is currently receiving (or has in the past 6 months) another treatment in combination with ibrutinib, such as anti-CD20 monoclonal antibody, BCL-2 antagonists such as venetoclax, or other novel treatments or chemotherapeutic agents. For clarification regarding specific medications not listed here, please discuss with the principal investigator
* COHORT 2: Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon) within 7 days of first dose of study drug and while on study
* COHORT 2: Concomitant use of a strong CYP3A inhibitor
* COHORT 2: Vaccinated with a live, attenuated vaccine within 4 weeks of registration
* COHORT 2: Patients with chronic liver disease and hepatic impairment meeting Child Pugh class B and C
* COHORT 2: History of stroke or intracranial hemorrhage within 6 months before registration
* COHORT 2: History of bleeding diathesis (e.g. hemophilia, von Willebrand disease)
* COHORT 2: Clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to registration
* COHORT 2: Chemotherapy for other malignancies
* COHORT 2: Concurrent systemic immunosuppressant therapy =< 21 days of the first dose of study drug with the exception of that which is part of the standard of care for COVID-19
* COHORT 2: Major surgery within 4 weeks of registration
* COHORT 2: Female subjects who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or within 1 month of last dose of study drug. Male subjects who plan to father a child while enrolled in this study or within 3 months after the last dose of study drug
* COHORT 2: Patients stopped ibrutinib >= 7 days prior to registration, for any reason
* COHORT 2: Patient is an active participant on investigational therapy through an Institutional Review Board (IRB) approved clinical trial for COVID-19 (NOTE: Participation through compassionate use protocol or expanded access is permitted)
* COHORT 2: At time of registration, the patient requires:

  * Endotracheal intubation and mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who require hospitalization for their COVID-19 disease or die (Cohort 1) | Up to 28 days after study registration
  Will calculate the proportion of patients who were outpatient at the time of study entry, and evaluate whether or not patients in this cohort required hospitalization associated with their coronavirus disease 2019 (COVID-19) infection.
Proportion of patients who require mechanical ventilation and/or die (Cohort 2) | Up to 28 days after study entry

SECONDARY OUTCOMES:
Rate of "flare phenomena" (Cohort I) | Up to 84 days
  Will characterize and calculate the proportion of patients who develop a "flare phenomenon" if ibrutinib is stopped. Will calculate corresponding 95% exact binomial confidence intervals for these outcomes. These will be graphically and quantitatively compared, where chi-square or Mantel-Haenszel-Cochran tests will be used to compare the numbers of patients who have the incident event of interest between treatment arms or other groups of interest.
Patient-reported health and symptom status (Cohort I) | Up to 84 days
  We will evaluate and characterize baseline status and changes in 8 primary COVID-19 related symptoms in these outpatient subjects: fever, loss of smell, cough, shortness of breath, fatigue, aching muscles, diarrhea, and decreased appetite. These will be assessed using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Resolution of symptoms will be defined as no fever, no loss of smell, and severity or frequency of the remaining six symptoms rated as 0 (none/never) or 1 (mild/rarely) on the PRO-CTCAE.
Patterns on ibrutinib therapy during COVID-19 infection (Cohort I) | Up to 84 days
  We will characterize and summarize overall and by B-cell histologic diagnosis whether or not patients suspend their ibrutinib therapy while in an outpatient setting during the first 28 days on study, and patterns of resumption of ibrutinib. Specifically, we will evaluate this outcome by assessing the number of days patients received ibrutinib in the first 28 days after enrollment on this trial.
Reasons for hospitalization (Cohort I) | Up to 84 days
Mortality (Cohort II) | Up to 84 days
Time to hospital discharge (Cohort II) | Up to 84 days
Intubation and oxygen supplementation (Cohort II) | Up to 84 days
  Will characterize and summarize the need for and duration of oxygen supplementation.
Incidence of "flare phenomena" (Cohort II) | Up to 84 days
Viral clearance | On days 15, 28, 42, and 56 after registration
  The proportions of patients who are documented as having viral clearance at the various time points will be summarized at each time point within each treatment arm. These proportions will be evaluated within as well as across the cohorts. Within each cohort, we will compare these rates at each of the time points using chi-square or Mantel-Haenszel-Cochran tests to assess differences between treatment arms or groups. Further, logistic regression models will be used to assess incidence of viral clearance and how treatment arm and other demographic and clinical factors affect the ability of patients to achieve viral clearance.
Development of COVID-19 antibodies | Up to 28 days
  The proportion of patients who are able to develop COVID-19 antibodies by days 15 and 28, defined as the number of patients who have a threshold level of detectable COVID-19 antibodies divided by the total number of patients in the specific cohort/arm.
Coagulopathy and thrombosis measures | Up to 28 days
Cytokine measures | Up to 84 days
  Will evaluate the baseline as well as change in plasma cytokines between treatment arms: IL-1beta, IL-1Ralpha, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL- IL-9, IL-10, IFNgamma, IP10, TNFalpha in longitudinal samples.
Immune subset measures | Up to 84 days
  Will evaluate the baseline as well as change in several immune cell subsets, including CD3 T cells, CD4 T-helper cells (and their subsets), CD8 T-suppressor cells (and their subsets), NK cells, B cells, and monocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer A Parikh, Principal Investigator — Academic and Community Cancer Research United
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States